CLINICAL TRIAL: NCT02650544
Title: Efficacy and Safety Analyses of Mirtazapine in the Treatment of Malignant Tumor Related Depression: A Phase II, Placebo-controlled, Randomized, Double-blinded Clinical Trial in Advanced Non-small Cell Lung Cancer Patients
Brief Title: Efficacy and Safety Analyses of Mirtazapine in NSCLC Patients With Depression
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, M.D. and Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MDES20150107
Record Dates: First submitted 2015-12-11; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Depression
Keywords: Carcinoma, Non-Small-Cell Lung; Depression; mirtazapine; patients health questionnaire (PHQ-9)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Depression | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mirtazapine (Experimental): Mirtazapine arm will be orally administered with mirtazapine 15mg, QD, consecutive medication for 8 weeks; along with palliative chemotherapy regimen decided by investigators.
  Interventions: Drug: Mirtazapine
- Placebo (Placebo Comparator): Placebo arm will be orally administered with placebo 15mg, QD, consecutive medication for 8 weeks; along with palliative chemotherapy regimen decided by investigators.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirtazapine — Patients in mirtazapine arm will be orally administered mirtazapine as an anti-depression therapy; along with palliative chemotherapy.
  Other Names: Treatment arm: mirtazapine administration
  Arms: mirtazapine
Drug: Placebo — Patients in placebo arm will be orally administered placebo; along with palliative chemotherapy.
  Other Names: Comparative arm: placebo administration
  Arms: Placebo

SUMMARY:
This is a phase II, placebo-controlled, randomized, double-blinded clinical trial. Study objective is to assess the efficacy and safety of mirtazapine in advanced NSCLC patients with malignant tumor related depression. Study hypothesis is that advanced NSCLC diagnosed with depression undertaking palliative chemotherapy with mirtazapine treatment for 8 weeks will have remarkable improvement in depression compared to baseline. Eligible advanced NSCLC Patients with PHQ-9 score ≥ 8, and undertaking palliative chemotherapy will be enrolled into this study. patients will be stratified (gender, age, Numerical Rating Scale score for cancer pain 0-3/4-6/7-10) randomized (1:1) into mirtazapine or placebo treatment. Patients in mirtazapine arm will be orally administered with mirtazapine 15mg, QD, consecutive medication for 8 weeks; along with palliative chemotherapy regimen decided by investigators. Patients in placebo arm will be orally administered with placebo 15mg, QD, consecutive medication for 8 weeks; along with palliative chemotherapy regimen decided by investigators. During the treatment, Patient health questionnaire (PHQ-9), Hamilton Depression Scale (HAMD-17) and European Organization for Research on Treatment of Cancer (EORTC) quality of life questionnaire-C30 (QLQ-C30) questionnaires will be collected at baseline, 3 weeks (d22) and 8 weeks (d57), or treatment discontinuation date due to depression deteriorated or suicidal tendency and behavior. Follow-up will last up to 4 weeks after treatment end with depression assessment (questionnaires every 2 weeks). Study endpoints: primary endpoint is the anti-depression efficacy (response rate). Response defined as the PHQ-9 or HAMD-17 questionnaire score decrease ≥ 50% compared with baseline level.

DETAILED DESCRIPTION:
Major depression prevail in patients with malignant tumor with an incident rate of 20% - 40%, 2-3 times more than the prevalence of population, especially high in patients with advanced solid tumor patients as 40% - 50.6%. National Comprehensive Cancer Network (NCCN) palliative care guideline recommended PHQ-9 as the diagnosis tool for depression, total scores ≥ 8 was considered the standard of malignant tumor related depression. Major depression had been proved related with malignant tumors, mirtazapine is the currently effective drug in anti-depression clinical therapy, have better tolerance and equal effect compared to Tricyclic antidepressants (TCAs) and 5-hydroxytryptamine (5-HT) or noradrenaline serotonin-norepinephrine reuptake inhibitors (NE-SNRIs).

This is a phase II, placebo-controlled, randomized, double-blinded clinical trial. Study objective is to assess the efficacy and safety of mirtazapine in advanced NSCLC patients with malignant tumor related depression. Study hypothesis is that advanced NSCLC diagnosed with depression undertaking palliative chemotherapy with mirtazapine treatment for 8 weeks will have remarkable improvement in depression compared to baseline. Palliative chemotherapy and mirtazapine have better efficacy, recovery rate, response duration, tolerance and quality of life improvement than palliative chemotherapy and placebo. Moreover, mirtazapine could improve patients' anxiety and chemotherapy related nausea and vomit.

Eligible advanced NSCLC Patients with PHQ-9 score ≥ 8, and undertaking palliative chemotherapy will be enrolled into this study. After baseline assessment (PHQ-9, HAMD-17 and EORTC QLQ-C30 questionnaires), 236 patients will be stratified (gender, age, NRS score for cancer pain 0-3/4-6/7-10) randomized (1:1) into mirtazapine or placebo treatment. Patients in mirtazapine arm will be orally administered with mirtazapine 15mg, QD, consecutive medication for 8 weeks; along with palliative chemotherapy regimen decided by investigators. Patients in placebo arm will be orally administered with placebo 15mg, QD, consecutive medication for 8 weeks; along with palliative chemotherapy regimen decided by investigators. During the treatment, PHQ-9, HAMD-17 and EORTC QLQ-C30 questionnaires will be collected at 3 weeks (d22) and 8 weeks (d57), or treatment discontinuation date due to depression deteriorated or suicidal tendency and behavior. Follow-up will last up to 4 weeks after treatment end with depression assessment (questionnaires every 2 weeks). If anti-depression therapy is not effective after 8 weeks treatment or treatment discontinuation, patients will be unblinded and receive other treatment according to investigators. Treatment end at 8 weeks.

Study endpoints: primary endpoint is the anti-depression efficacy (response rate). Response defined as the PHQ-9 or HAMD-17 questionnaire score decrease ≥ 50% compared with baseline level. Secondary endpoints included: 1.recovery rate, recovery defined as the PHQ-9 score less than 8 points. 2. Response duration, defined as the time period from treatment response to regression recurrence (PHQ-9 score ascending above baseline level). 3. Quality of life improvement, define as the best quality of life score minus baseline level. 4. Compliance to anti-depression therapy, defined as the medication count at each follow-up time points.

ELIGIBILITY:
Inclusion Criteria:

* Pathology confirmed non-small cell lung cancer, undertaking palliative chemotherapy
* Age above 18 years old
* PHQ-9 score ≥ 8 points at baseline assessment
* Eastern Cooperative Oncology Group (ECOG) performance score 0 -2
* Orally administration of drugs without difficulties
* Eligible bone marrow function, liver and kidney function for chemotherapy
* Pregnancy test negative in 7 days for women of child-bearing age; willing to take contraception measures.
* Signed Informed consent form (ICF)

Exclusion Criteria:

* Clinical diagnosis of depression before advanced NSCLC confirmed
* Suicide tendency or behavior
* Mania in past medical history
* Received surgery or radiation therapy in 4 weeks
* Central nervous system (CNS) metastasis or spinal compression; except no symptoms and with no cortical hormonotherapy in 4 weeks.
* Systemically treatment with psychotropic medications, antihistamines drugs, antibiotics, cortical hormone therapy, antiepileptic drugs, immunosuppressive agents or other drugs might affect treatment in 4 weeks; or locally used of these drug in 2 weeks.
* AST or ALT ≥ 2.5 ULN without liver metastasis; or ≥ 5 ULN with liver metastasis.
* Serum creatinine ≥ 2 mg/dl
* Residual toxicity event ≥ CTCAE grade 2, except peripheral neurotoxicities.
* Any severe or uncontrolled systemic diseases judged by investigators.
* Any contraindication of mirtazapine.

Exclusion Criteria:

* Invalid subject after randomization
* Major protocol violations judged by investigators.
* Poor compliance
* Intolerable adverse events
* Subject withdraw ICF
* Any pregnancy events
* No clinical benefits due to clinical adverse events, laboratory abnormalities or other medical conditions
* Other reasons of treatment discontinuation judged by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants responded to treatment. | baseline, and 3 weeks (d22), and 8 weeks (d57), and follow-up (d71, d85)
  Using PHQ-9 or HAMD-17 questionnaire to assess the change of depression scores at the time points above. The measure unit is questionnaire score point, remain the same at every time points. And to calculate response number of patients (patients had 50% percent of depression questionnaire score points reduction compared to baseline after treatment initiation) and recovery number of patients (patients had PHQ-9 score less than 8 points PHQ-9 score less than 8 points during the treatment).

SECONDARY OUTCOMES:
Response duration | From date of randomization until the date of first documented regression recurrence, assessed up to 12 weeks"
  Regression recurrence defined as PHQ-9 score ascending above baseline level.
Number of participants had quality of life improvement | baseline, and 3 weeks (d22), and 8 weeks (d57), and follow-up (d71, d85)
  Using EORTC QLQ-C30 (V3.0) to assess the quality of life change at the time points above. The measure unit is questionnaire score point, remain the same at every time points. And to calculate improved number of patients (patients had quality of life questionnaire score points gained compared to baseline after treatment initiation)

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, professor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center of Sun-Yat Sen University (CCSYSU), Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reddy MS. Depression: the disorder and the burden. Indian J Psychol Med. 2010 Jan;32(1):1-2. doi: 10.4103/0253-7176.70510. No abstract available. PMID 21799550
- [Background] Sharpe M, Walker J, Holm Hansen C, Martin P, Symeonides S, Gourley C, Wall L, Weller D, Murray G; SMaRT (Symptom Management Research Trials) Oncology-2 Team. Integrated collaborative care for comorbid major depression in patients with cancer (SMaRT Oncology-2): a multicentre randomised controlled effectiveness trial. Lancet. 2014 Sep 20;384(9948):1099-108. doi: 10.1016/S0140-6736(14)61231-9. Epub 2014 Aug 27. PMID 25175478
- [Background] Stafford L, Judd F, Gibson P, Komiti A, Mann GB, Quinn M. Anxiety and depression symptoms in the 2 years following diagnosis of breast or gynaecologic cancer: prevalence, course and determinants of outcome. Support Care Cancer. 2015 Aug;23(8):2215-24. doi: 10.1007/s00520-014-2571-y. Epub 2015 Jan 6. PMID 25559036
- [Background] Walker J, Hansen CH, Martin P, Symeonides S, Gourley C, Wall L, Weller D, Murray G, Sharpe M; SMaRT (Symptom Management Research Trials) Oncology-3 Team. Integrated collaborative care for major depression comorbid with a poor prognosis cancer (SMaRT Oncology-3): a multicentre randomised controlled trial in patients with lung cancer. Lancet Oncol. 2014 Sep;15(10):1168-76. doi: 10.1016/S1470-2045(14)70343-2. Epub 2014 Aug 27. PMID 25175097
- [Background] Rodin G. Effective treatment for depression in patients with cancer. Lancet. 2014 Sep 20;384(9948):1076-8. doi: 10.1016/S0140-6736(14)61342-8. Epub 2014 Aug 28. No abstract available. PMID 25175951
- [Background] Andersen BL, Rowland JH, Somerfield MR. Screening, assessment, and care of anxiety and depressive symptoms in adults with cancer: an american society of clinical oncology guideline adaptation. J Oncol Pract. 2015 Mar;11(2):133-4. doi: 10.1200/JOP.2014.002311. Epub 2014 Dec 16. No abstract available. PMID 25515721
- [Background] Amini H, Aghayan S, Jalili SA, Akhondzadeh S, Yahyazadeh O, Pakravan-Nejad M. Comparison of mirtazapine and fluoxetine in the treatment of major depressive disorder: a double-blind, randomized trial. J Clin Pharm Ther. 2005 Apr;30(2):133-8. doi: 10.1111/j.1365-2710.2004.00585.x. PMID 15811165
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Spiegel D. Minding the body: psychotherapy and cancer survival. Br J Health Psychol. 2014 Sep;19(3):465-85. doi: 10.1111/bjhp.12061. Epub 2013 Aug 26. PMID 23980690
- [Background] Massie MJ. Prevalence of depression in patients with cancer. J Natl Cancer Inst Monogr. 2004;(32):57-71. doi: 10.1093/jncimonographs/lgh014. PMID 15263042
- [Background] Hopwood P, Stephens RJ. Depression in patients with lung cancer: prevalence and risk factors derived from quality-of-life data. J Clin Oncol. 2000 Feb;18(4):893-903. doi: 10.1200/JCO.2000.18.4.893. PMID 10673533
- [Background] Arrieta O, Angulo LP, Nunez-Valencia C, Dorantes-Gallareta Y, Macedo EO, Martinez-Lopez D, Alvarado S, Corona-Cruz JF, Onate-Ocana LF. Association of depression and anxiety on quality of life, treatment adherence, and prognosis in patients with advanced non-small cell lung cancer. Ann Surg Oncol. 2013 Jun;20(6):1941-8. doi: 10.1245/s10434-012-2793-5. Epub 2012 Dec 22. PMID 23263699
- [Background] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Background] de Souza BF, de Moraes JA, Inocenti A, dos Santos MA, Silva AE, Miasso AI. Women with breast cancer taking chemotherapy: depression symptoms and treatment adherence. Rev Lat Am Enfermagem. 2014 Oct;22(5):866-73. doi: 10.1590/0104-1169.3564.2491. PMID 25493684
- [Background] Badr H, Shen MJ. Pain catastrophizing, pain intensity, and dyadic adjustment influence patient and partner depression in metastatic breast cancer. Clin J Pain. 2014 Nov;30(11):923-33. doi: 10.1097/AJP.0000000000000058. PMID 24402001
- [Background] Lee Y, Lin PY, Chien CY, Fang FM. Prevalence and risk factors of depressive disorder in caregivers of patients with head and neck cancer. Psychooncology. 2015 Feb;24(2):155-61. doi: 10.1002/pon.3619. Epub 2014 Jul 10. PMID 25045052
- [Background] Theobald DE, Kirsh KL, Holtsclaw E, Donaghy K, Passik SD. An open-label, crossover trial of mirtazapine (15 and 30 mg) in cancer patients with pain and other distressing symptoms. J Pain Symptom Manage. 2002 May;23(5):442-7. doi: 10.1016/s0885-3924(02)00381-0. PMID 12007762
- [Background] Burrows GD, Kremer CM. Mirtazapine: clinical advantages in the treatment of depression. J Clin Psychopharmacol. 1997 Apr;17 Suppl 1:34S-39S. doi: 10.1097/00004714-199704001-00005. PMID 9090576
- [Background] Anttila SA, Leinonen EV. A review of the pharmacological and clinical profile of mirtazapine. CNS Drug Rev. 2001 Fall;7(3):249-64. doi: 10.1111/j.1527-3458.2001.tb00198.x. PMID 11607047
- [Background] Ito T, Okubo Y, Roth A. [Efficacy of mirtazapine for appetite loss and nausea of the cancer patient--from clinical experience in Memorial Sloan-Kettering Cancer Center]. Gan To Kagaku Ryoho. 2009 Apr;36(4):623-6. Japanese. PMID 19381036 (Retraction: PMID 19891088 Ito T, Sato H. Gan To Kagaku Ryoho. 2009 Oct;36(10):1779)
- [Background] Puzantian T. Mirtazapine, an antidepressant. Am J Health Syst Pharm. 1998 Jan 1;55(1):44-9. doi: 10.1093/ajhp/55.1.44. PMID 9437474
- [Background] Sanacora G, Treccani G, Popoli M. Towards a glutamate hypothesis of depression: an emerging frontier of neuropsychopharmacology for mood disorders. Neuropharmacology. 2012 Jan;62(1):63-77. doi: 10.1016/j.neuropharm.2011.07.036. Epub 2011 Aug 3. PMID 21827775
- [Background] Popoli M, Yan Z, McEwen BS, Sanacora G. The stressed synapse: the impact of stress and glucocorticoids on glutamate transmission. Nat Rev Neurosci. 2011 Nov 30;13(1):22-37. doi: 10.1038/nrn3138. PMID 22127301
- [Background] Huntzinger E, Izaurralde E. Gene silencing by microRNAs: contributions of translational repression and mRNA decay. Nat Rev Genet. 2011 Feb;12(2):99-110. doi: 10.1038/nrg2936. PMID 21245828
- [Background] Zeng LH, Rensing NR, Wong M. Developing Antiepileptogenic Drugs for Acquired Epilepsy: Targeting the Mammalian Target of Rapamycin (mTOR) Pathway. Mol Cell Pharmacol. 2009 Jan 1;1(3):124-129. doi: 10.4255/mcpharmacol.09.16. PMID 20419051
- [Background] Smalheiser NR, Lugli G, Rizavi HS, Torvik VI, Turecki G, Dwivedi Y. MicroRNA expression is down-regulated and reorganized in prefrontal cortex of depressed suicide subjects. PLoS One. 2012;7(3):e33201. doi: 10.1371/journal.pone.0033201. Epub 2012 Mar 9. PMID 22427989
- [Background] Baudry A, Mouillet-Richard S, Schneider B, Launay JM, Kellermann O. miR-16 targets the serotonin transporter: a new facet for adaptive responses to antidepressants. Science. 2010 Sep 17;329(5998):1537-41. doi: 10.1126/science.1193692. PMID 20847275
- [Background] Issler O, Haramati S, Paul ED, Maeno H, Navon I, Zwang R, Gil S, Mayberg HS, Dunlop BW, Menke A, Awatramani R, Binder EB, Deneris ES, Lowry CA, Chen A. MicroRNA 135 is essential for chronic stress resiliency, antidepressant efficacy, and intact serotonergic activity. Neuron. 2014 Jul 16;83(2):344-360. doi: 10.1016/j.neuron.2014.05.042. Epub 2014 Jun 19. PMID 24952960
- [Background] Bocchio-Chiavetto L, Maffioletti E, Bettinsoli P, Giovannini C, Bignotti S, Tardito D, Corrada D, Milanesi L, Gennarelli M. Blood microRNA changes in depressed patients during antidepressant treatment. Eur Neuropsychopharmacol. 2013 Jul;23(7):602-11. doi: 10.1016/j.euroneuro.2012.06.013. Epub 2012 Aug 25. PMID 22925464
- [Background] Lotrich FE. Inflammatory cytokine-associated depression. Brain Res. 2015 Aug 18;1617:113-25. doi: 10.1016/j.brainres.2014.06.032. Epub 2014 Jul 5. PMID 25003554